CLINICAL TRIAL: NCT06155084
Title: A Phase I/II Open-Label Study to Assess the Safety, Pharmacokinetics, and Antitumor Activity of Oral HP518 in Patients With Metastatic Castration-Resistant Prostate Cancer in China
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Anti-Tumor Activity of Oral HP518 in mCRPC Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hinova Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HP518-01-01-03
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 - Dose Escalation, 400mg/d (Cohort1) (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: HP518 - Dose Escalation
- Part 1 - Dose Escalation 500mg/d (Cohort 2) (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: HP518 - Dose Escalation
- Part 2 - Dose Expansion Oral tablet(s) (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: HP518 -Dose Expansion

INTERVENTIONS:
Drug: HP518 - Dose Escalation — Part 1: Dose escalation Daily oral dosage with the prescribed dose level based on Cohort
  Other Names: Part 1 - Dose Escalation
  Arms: Part 1 - Dose Escalation, 400mg/d (Cohort1)
Drug: HP518 - Dose Escalation — Part 1: Dose escalation Daily oral dosage with the prescribed dose level based on Cohort
  Other Names: Part 1 - Dose Escalation
  Arms: Part 1 - Dose Escalation 500mg/d (Cohort 2)
Drug: HP518 -Dose Expansion — Part 2: Dose expansion Daily oral dosage with the highest dose with acceptable toxicity (RP2D) based on data from Part 1.
  Other Names: Part 2 - Dose Expansion Oral tablet(s)
  Arms: Part 2 - Dose Expansion Oral tablet(s)

SUMMARY:
The overall objective of this Phase 1 study is to evaluate the safety, PK,and anti-tumor activity of daily oral dosing with HP518,selecting the RP2D of HP518 based on assessments of patients with progressive mCRPC in dose-escalation phase

DETAILED DESCRIPTION:
This First in Human dose escalation and expansion study of HP518 in patients with progressive mCRPC after NHA and chemotherapy is being conducted not only to evaluate the safety and tolerability of orally administered HP518, but also to provide preliminary efficacy for the reference of future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age ≥18
2. Patients with androgen receptor (AR) ligand binding domain (LBD) activation mutations (the dose expansion part of stage II)
3. Has histologically confirmed adenocarcinoma of the prostate, but there are no known significant neuroendocrine differentiation or small cell characteristics.
4. Has metastatic disease documented by 2 or more bone lesions by bone scan or soft tissue disease progression observed by CT/MRI at the beginning of study.
5. the progression of the disease after receiving at least one new endocrine therapy and progressing with at least first-line chemotherapy.
6. Must have recovered from toxicities related to any prior treatments
7. Ongoing ADT with LHRH agonist/antagonist therapy or history of bilateral orchiectomy.
8. ECOG performance status score of 0 to 1.

Exclusion Criteria:

1. Combination of research or commercially available drugs targeting AR
2. Has had any other anticancer treatments, including immunotherapy, chemotherapy, or radiotherapy (eg, 177LuPSMA-617, radium 223, PARP inhibitor) within 4 weeks prior to the first dose of HP518.
3. Has gastrointestinal disorder affecting absorption (e.g., gastrectomy).
4. Has significant cardiovascular disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidences of Protocol-defined DLT during the DLT assessment period , characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drugorally administered HP518 (Part 1) | 28 DAYS
  To evaluate the safety and tolerability and determine the MTD and the RP2D of orally administered HP518 (Part 1)
Incidence of Treatment-Emergent Adverse Events characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness | Through study completion, an average of 1 year
  To evaluate the safety of orally administered HP518 (Part 1)
Incidence of laboratory abnormalities, characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing | Through study completion, an average of 1 year
  To evaluate the safety of orally administered HP518 (Part 1)
Incidence of vital signs abnormalities characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing | Through study completion, an average of 1 year
  To evaluate the safety of orally administered HP518 (Part 1)
Incidence of ECG (PR, QRS, QT, and QTcF intervals) abnormalities characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing | Through study completion, an average of 1 year
  To evaluate the safety of orally administered HP518 (Part 1)
PSA50 response rate | 12 weeks
  Proportion of patients showing a PSA decline by ≥50% between baseline and Week 12 of dosing with HP518.

SECONDARY OUTCOMES:
area under the concentration-time curve (AUC) | 12 weeks
  Assessment of pharmacokinetic parameters of HP518
Maximum concentration (Cmax) | 12 weeks
  Assessment of pharmacokinetic parameters of HP518
Time to maximum concentration (Tmax) | 12 weeks
  Assessment of pharmacokinetic parameters of HP518
Apparent terminal elimination half-life (T1/2) | 12 weeks
  Assessment of pharmacokinetic parameters of HP518
apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | 12 weeks
  Assessment of pharmacokinetic parameters of HP518
oral clearance (CL/F) | 12 weeks
  Assessment of pharmacokinetic parameters of HP518
According to PCWG3 | 8 weeks
  evaluate PSA50 response rate: PSA decline by≥50% between baseline and 4 weeks/8 weeks/12 weeks( only Part 1) of dosing with HP518
According to PCWG3, evaluate time to PSA progression | Through study completion, an average of 1 year
  PCWG3 definition: PSA increase >25% and >2 ng/mL above nadir, confirmed by progression at 2 time points at least 3 weeks apart) nadir, confirmed by progression at 2 time points at least 3 weeks apart)
Time to radiographic progression by investigator PCWG3 definition | Through study completion, an average of 1 year
  using the RECIST v1.1 and PCWG3 definition
Evaluate the modified best overall response mBOR by investigator | Through study completion, an average of 1 year
  According to RECIST (version 1.1) and PCWG3
analyze the efficacy of patients with different AR phenotypes(Part 2) | Through study completion, an average of 1 year
  According to genetic testing results

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - The Second Hospital Of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Xiamen Univeristy, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital Of Guizhou Medical University, Guiyang, Guizhou
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital Of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital Of Xi'An Jiaotong Univeristy, Xi’an, Shanxi
  - Sichuan Academy of Medical Science & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital Of Sichuan University, Chengdu, Sichuan
  - The Affiliated Hospital Of Southwest Medical University, Luzhou, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - The Second Affiliated Hospital Of Kunming Medical University, Kunming, Yunnan
  - The Affiliated Hospital Of School Of Medicine Of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No